CLINICAL TRIAL: NCT03122535
Title: 70 Versus 110 Degrees Side-cut Angles in Femtosecond Laser-assisted in Situ Keratomileusis
Brief Title: 70 vs 110 Degree Side-cut Angles in Femtosecond LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Mark Mifflin, Clinical Professor, Ophthalmology/Visual Sciences, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB 74858
Record Dates: First submitted 2017-02-18; First posted 2017-04-20 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Operative Incision
Keywords: Femtosecond LASIK (FS--LASIK); Visual acuity; Refractive errors; Side-cut angles
MeSH Terms: conditions — Surgical Wound; Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Masking Description: Each participant will be masked as to which angle of cut is used in which eye. Each patient will receive a 70 degree cut in one eye and a 110 degree cut in the fellow eye
Oversight: Data Monitoring Committee: No

ARMS (2):
- FS-LASIK 70 degree side-cut angle (Active Comparator): Each patient will be masked as to which angle of cut is used in which eye. Each patient will receive a 70 degree cut in one eye and a 110 degree cut in the fellow eye.
  Interventions: Device: FS-LASIK 70 degree side-cut angle; Device: FS-LASIK 110 degree side-cut angle
- FS-LASIK 110 degree side-cut angle (Active Comparator): Each patient will be masked as to which angle of cut is used in which eye. Each patient will receive a 70 degree cut in one eye and a 110 degree cut in the fellow eye.
  Interventions: Device: FS-LASIK 70 degree side-cut angle; Device: FS-LASIK 110 degree side-cut angle

INTERVENTIONS:
Device: FS-LASIK 70 degree side-cut angle — FS-LASIK surgical procedures will be performed according to the surgeons' standard practices. Patient will be masked as to the treatment they receive in either eye so as not to influence their subjective responses and visual measurements. Patients will be discontinued from the study if, on the day of surgery, both eyes cannot be randomized and operated as per protocol.
Device: FS-LASIK 110 degree side-cut angle — FS-LASIK surgical procedures will be performed according to the surgeons' standard practices. Patient will be masked as to the treatment they receive in either eye so as not to influence their subjective responses and visual measurements. Patients will be discontinued from the study if, on the day of surgery, both eyes cannot be randomized and operated as per protocol.

SUMMARY:
The purpose of this study is to compare 70 and 110 degree side-cut angles on the same patient undergoing Femtosecond Laser-assisted in Situ Keratomileusis (FS-LASIK).

DETAILED DESCRIPTION:
LASIK has become the preferred corneal procedure to correct certain refractive errors. One of the major advancements in LASIK has been the introduction of Femtosecond Laser technology for flap creation. Several studies have compared microkeratome and femtosecond laser technology, showing superior accuracy and precision of flap dimensions in the latter.

The Femtosecond Laser technology provides different parameters and settings that can be changed according to the surgeon's preference. One of such parameters is the side-cut angle. Some of the most common side-cut angles used today include 45, 70, 90, and 110 degrees. Previous studies have reported on the visual outcomes of side-cut angles, but head to head comparisons are lacking. Currently, there are no studies comparing the safety and efficacy of the 70 and 110 side-cut angles in FS-LASIK. Information regarding the outcomes and complication rates between these side-cut angles will provide an objective measure that can be used when deciding which one is more suitable in FS-LASIK.

One angle will be performed on the right eye and the other on the left eye. The study will evaluate uncorrected visual acuity, best corrected visual acuity, intraoperative, and postoperative complications. Performing different side-cut angles on the same individual will allow a direct comparison of outcomes, minimizing confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are deemed suitable candidates for bilateral LASIK will be considered eligible for participation in this study. Correction will be distance for both eyes.

Exclusion Criteria:

* Selection will be consistent with current standard of care. Any patient that is not a suitable candidate for LASIK will not be included.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Mifflin, MD, Principal Investigator — University of Utah Moran Eye Center
Locations (1):
- University of Utah John A. Moran Eye Center - Midvalley Location, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | FS-LASIK 70 Degree Side-cut Angle | FS-LASIK 110 Degree Side-cut Angle
Started | 115; 115 Eyes | 115; 115 Eyes
3 Months | 92; 92 Eyes | 92; 92 Eyes
12 Months | 42; 42 Eyes | 42; 42 Eyes
Completed | 42; 42 Eyes | 42; 42 Eyes
Not Completed | 73; 73 Eyes | 73; 73 Eyes
Not completed — Lost to Follow-up | 68 | 68
Not completed — Physician Decision | 3 | 3
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Each patient will be masked as to which angle of cut is used in which eye. Each patient will receive a 70 degree cut in one eye and a 110 degree cut in the fellow eye.
  FS-LASIK 70 degree side-cut angle: FS-LASIK surgical procedures will be performed according to the surgeons' standard practices. Patient will be masked as to the treatment they receive in either eye so as not to influence their subjective responses and visual measurements. Patients will be discontinued from the study if, on the day of surgery, both eyes cannot be randomized and operated as per protocol.
  FS-LASIK 110 degree side-cut angle: FS-LASIK surgical procedures will be performed according to the surgeons' standard practices. Patient will be masked as to the treatment they receive in either eye so as not to influence their subjective responses and visual measurements. Patients will be discontinued from the study if, on the day of surgery, both eyes cannot be randomized and operated as per protocol.
Arm/Group | All Participants
Number analyzed (Participants) | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 115
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.96 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 93
  More than one race | 5
  Unknown or Not Reported | 12

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Visual Acuity at One Year
Description: Vision testing without correction, both eyes using Snellen Eye chart
Time Frame: one year
Population: This is a contralateral eye study of 115 subjects, each with one eye randomized to the two study groups.
Measure: Mean (Standard Deviation); unit: logMAR Visual Acuity
Arm/Group | FS-LASIK 70 Degree Side-cut Angle | FS-LASIK 110 Degree Side-cut Angle
Number analyzed (Participants) | 115 | 115
logMAR Visual Acuity | -0.082 (0.065) | -0.094 (0.072)

2. Secondary Outcome: Best Corrected Visual Acuity at Year One
Description: Vision testing with correction, both eyes using Snellen Eye chart
Time Frame: one year
Measure: Mean (Standard Deviation); unit: logMAR Visual Acuity
Arm/Group | FS-LASIK 70 Degree Side-cut Angle | FS-LASIK 110 Degree Side-cut Angle
Number analyzed (Participants) | 115 | 115
logMAR Visual Acuity | -0.109 (0.066) | -0.116 (0.060)

ADVERSE EVENTS:
Time Frame: 1 year
Description: No risk for mortality from treatment
Arm/Group | FS-LASIK 70 Degree Side-cut Angle | FS-LASIK 110 Degree Side-cut Angle
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/115
Other Adverse Events (participants affected / at risk) | 2/115 | 2/115
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS-LASIK 70 Degree Side-cut Angle (N=115) | FS-LASIK 110 Degree Side-cut Angle (N=115)
Enhancement Needed (Surgical and medical procedures) | 2 (2) | 2 (2) — Eye needed an enhancement as uncorrected visual acuity was deemed unacceptable and needed to be improved with additional treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT03122535/Prot_SAP_000.pdf